CLINICAL TRIAL: NCT05487001
Title: Analgesic Effect of Dexamethasone as a Perineural Adjuvant for Continuous Femoral Nerve Block After Total Knee Arthroplasty: a Prospective Randomized Placebo-controlled Trial
Brief Title: Perineural Dexamethasone for Continuous Femoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Myoung Hwa Kim, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3-2022-0230
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexamethasone group (Experimental): a iliopsoas plane block before surgery
  Interventions: Procedure: dexamethasone group
- sham group (Sham Comparator): sham block before surgery
  Interventions: Procedure: sham group

INTERVENTIONS:
Procedure: dexamethasone group — 1) Arm l (dexamethasone group) Ultrasound-guided femoral nerve block with 1% lidocaine 15 ml after the end of surgery Postoperative femoral nerve patient controlled analgesia
  * Total volume 250 ml (0.375% ropivacaine 60 ml + normal saline 188 ml + dexamethasone 10 mg (2 ml))
  * Basal rate 4 mL/hr, Bolus volume 2 mL, Lock-out time 15 min
  Arms: dexamethasone group
Procedure: sham group — 2) Arm ll (sham group) Ultrasound-guided femoral nerve block with 1% lidocaine 15 ml after the end of surgery Postoperative femoral nerve patient controlled analgesia
  * Total volume 250 ml (0.375% ropivacaine 60 ml + normal saline 190 ml
  * Basal rate 4 mL/hr, Bolus volume 2 mL, Lock-out time 15 min
  Arms: sham group

SUMMARY:
An alternative to improve the quality of postoperative analgesia is to use various perineural adjuvants applicable to peripheral nerve block along with local anesthetics to increase the analgesic effect. Dexamethasone is a strong and long-acting corticosteroid, which reduces postoperative nausea and vomiting and increases the duration of nerve blockade. Most of the existing clinical studies compared the analgesic effect with the placebo group after adding an adjuvant in a single shot nerve block, and there were very few cases of comparing the analgesic effect with the placebo group after adding the adjuvant in peripheral nerve block through continuous catheter infusion. Therefore, we designed this study to investigate whether the use of dexamethasone as a peripheral adjuvant for continuous femoral nerve block has a better pain and recovery profile.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19 years of age or older who are expected to undergo unilateral hip arthroplasty
2. ASA PS 1-3

Exclusion Criteria:

1. Revision total hip arthroplasty
2. Allergy to drugs used in the study
3. Patients with moderate or more hepatic impairment (AST/ALT is more than 2.5 times the upper limit of normal)
4. Estimated glomerular filtration rate < 30 mL/min/1.73m2
5. Opioid dependence
6. Prolongation of PT and aPTT more than twice the upper limit of normal
7. Pre-existing neurological or anatomical disorders of the lower extremities
8. Serious psychiatric disorders

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Maximum Numeric rating scale pain score at movement | within postoperative day 2
  Pain intensity at movement will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) postoperative 1 hour, postoperative 6 hours, postoperative day 1, postoperative day 2. Maximum Numeric rating scale pain score was determined based on highest score among repeated assessment of surgical site pain severity postoperatively.

SECONDARY OUTCOMES:
Numeric rating scale pain score at rest | up to postoperative day 2
  Pain intensity at rest will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) postoperative 1 hour, postoperative 6 hours, postoperative day 1, postoperative day 2.
Numeric rating scale pain score at movement | up to postoperative day 2
  Pain intensity during 45-degree passive flexion of the hip with the ipsilateral knee flexed naturally will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) postoperative 1 hour, postoperative 6 hours, postoperative day 1, postoperative day 2.
Postoperative opioid consumption | up to postoperative day 2
  morphine equivalent dose

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No